CLINICAL TRIAL: NCT04230902
Title: A Prospective Randomized Comparative Clinical Trial Evaluating the Effects of Autologous Microfractured Adipose Tissue (α MAT) Versus Steroid Injection in Knee Osteoarthritis (STα MAT-knee Study)
Brief Title: Effects of α MAT Versus Steroid Injection in Knee Osteoarthritis (STα MAT-knee Study)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Hasan Baydoun, Clinical Instructor, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIO-2017-0440
Record Dates: First submitted 2019-01-29; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Knee Osteoarthritis
Keywords: mesenchymal stem cell; corticosteroid; adipose stem cell; MRI; pain; Knee
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Adrenal Cortex Hormones; Steroids

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lipogems (Experimental): The cases assigned to this group will be injected intra-articularly with Lipogems®. The patients will undergo harvesting of their own adipose tissue for aMAT then this aMAT will be injected intra-articularly in the knee. It will be administered once at the baseline visit of the study.
  Interventions: Biological: Microfragmented Adipose Tissue Transplant
- Steroid (Active Comparator): The cases assigned to this group will be injected intra-articularly in the knee with corticosteroids. No extra preparation of any type is necessary in this case. It will be administered once at the baseline visit of the study.
  Interventions: Drug: Corticosteroid injection

INTERVENTIONS:
Biological: Microfragmented Adipose Tissue Transplant — Autologous Microfragmented Adipose Tissue derived using Lipogems® Kit
  Other Names: aMAT
  Arms: Lipogems
Drug: Corticosteroid injection — intra-articular knee injection of corticosteroid
  Other Names: steroid
  Arms: Steroid

SUMMARY:
Knee Osteoarthritis (OA) is a common degenerative knee condition of the knee which is treated symptomatically. Knee cartilage tissue has little regenerative ability With the developments in regenerative medicine, stem cells might also be used in knee OA. Recently, adipose tissue has been identified as means for autologous mesenchymal stem cells (aMAT) using non-enzymatic method. Lipogems® is FDA-approved closed-system and directly producing ready-to-use aMAT. Some observational studies showed its potential in knee chondropathy. With no clinical trial done as yet, the investigators will hereby study the comparative efficacy of corticosteroid (current practice) versus Lipogems® in patients with knee OA. The knee MRI changes, clinical and patient-based outcomes will compared between baseline and throughout till 6 months after treatment. This study aims to show the comparative efficacy of Lipogems® as compared to corticosteroid in knee OA patients and to demonstrate its cartilage regeneration potential, which will ultimately deter surgery.

DETAILED DESCRIPTION:
Knee Osteoarthritis (OA) is a common degenerative condition of the knee. Its current management is symptomatic. These patients might eventually need total knee arthroplasty (TKA). With the developments in regenerative medicine, stem cell has been suggested as means to regenerate the knee cartilage tissue which otherwise has little regenerative ability. Initially, stem cells were obtained from bone marrow cells; however, now they can also be obtained from adipose tissue through liposuction. With developments of less invasive liposuction techniques, adipose tissue has been identified as means for autologous mesenchymal stem cells (aMAT). There are two ways of obtaining aMAT form adipose tissue: enzymatic, which has controversies related to Good Manufacturing Practice and low yield, and non-enzymatic method which was recently further developed to a closed-system and directly ready-to-use aMAT producing Lipogems®. Lipogems® is FDA-approved for several applications including orthopedic use. A couple of case reports and cohort studies showed its potential use in knee chondropathy. Until now, no clinical trials compared its effect to the knee OA standard of care which is the intra-articular corticosteroid injection. Here, the investigators will study the comparative efficacy of corticosteroid versus Lipogems® in patients with knee OA.

This randomized clinical trial will include 48 patients with symptomatic knee OA ≥ 45 years old with no contraindication of corticosteroid and/or Lipogems® use. These patients will be divided equally into two groups: group S who will receive intra-articular corticosteroid knee injection and group L whose aMAT will be harvested using Lipogems® and be injected intra-articularly. The knee pain, clinical parameters, and patient-related outcome measures (knee injury and osteoarthritis outcome score and Lipogems® Questionnaire-knee) will be assessed at baseline, 2-week, 6-week, 3-month, and 6-month. Also, knee MRI will be done at baseline and 6-months to visualize any changes (MRI Osteoarthritis knee score). These outcomes will be evaluated over the 6-month period and the difference between baseline and follow-up will be compared between the two groups.

This study aims to show the comparative efficacy of Lipogems® as compared to corticosteroid in knee OA patients and to demonstrate its cartilage regeneration potential, which will ultimately deter surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are ≥ 45 years old
* Symptomatic knee OA defined as symptoms of knee pain and/or decreased range of motion (ROM)
* Classified radiographically as having Grade 2 or 3 Knee OA
* Failure of 3-months conservative management (NSAIDs and Physical therapy)

Exclusion Criteria:

* Patients < 45 years old
* Pregnant or breastfeeding women
* Cancer patients
* Rheumatoid arthritis patients
* Patients having any autoimmune disease affecting the joint
* Patients who have had hyaluronic acid injection <1 year ago
* Patients who have undergone lower extremity surgery or trauma on the same side
* Hypersensitivity to methylprednisolone (Depo-Medrol®)or any of its components, lidocaine/xylocaine or any of its components, and any of the ingredients of Lipogems® injection kit
* Patients with acute systemic or local infection
* Patients on anticoagulants (warfarin, coumadin, heparin, Xeralto, or Plavix)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-03-04 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Comparing the total pain score pre- and post-injection differences between the two arms | 6 months
  The difference in total pain scores (using numerical rating scale) between the baseline visit (prior to injection) and 6 months after injection will be obtained for each arm. And these differences will be compared between Lipogems and Steroid arms using t-test to assess the effect of each injection type on pain severity
Comparing MOAKS pre-and post-injection differences between the two arms | 6 months
  The difference in MOAKS values (MRI Osteoarthritis Knee Score) between the baseline visit (prior to injection) and 6 months after injection will be obtained for each arm. And these differences will be compared between Lipogems and Steroid arms using t-test to assess the anatomic effects of each injection type.

SECONDARY OUTCOMES:
Clinical outcomes-extension | 6 months (at 0weeks, 2weeks, 6weeks, 3months, and 6months)
  The extension lag (in degrees by clinical exam) as assessed by the clinician at baseline (0, pre-injection) and each visit (2 weeks, 6weeks, 3months, and 6months) will be noted and compared between the two arms at each visit timepoint
Clinical outcomes-flexion | 6 months (at 0weeks, 2weeks, 6weeks, 3months, and 6months)
  The flexion range (in degrees by clinical exam) as assessed by the clinician at baseline (0, pre-injection) and each visit (2 weeks, 6weeks, 3months, and 6months) will be noted and compared between the two arms at each visit timepoint
Clinical outcomes-stability | 6 months (at 0weeks, 2weeks, 6weeks, 3months, and 6months)
  The knee stability (presence/absence) results as assessed by the clinician at baseline (0, pre-injection) and each visit (2 weeks, 6weeks, 3months, and 6months) will be noted and compared between the two arms at each visit timepoint
Cartilage thickness | 6 months (at 0weeks & 6months)
  Comparing the average difference in thickness of the knee cartilage (in mm), measured on MR image, between the two arms between baseline and 6 months.
Patient-based outcomes | 6 months (at 0weeks, 2weeks, 6weeks, 3months, and 6months)
  The difference scores of patient-based outcome questionnaires (Lipogems® Questionnaire-Knee, and Knee injury and Osteoarthritis Outcome Score or KOOS) between baseline and post-injection follow-ups (2weeks, 6 weeks, 3months, 6 months) will be measured. These difference in scores will be compared between the two arms.
Pain score-other follow-ups | 3 months (at 0weeks, 2weeks, 6weeks, 3months)
  The difference in pain scores (numerical rating scale) between the baseline visit (prior to injection) and at each follow-up visit (2 weeks, 6 weeks, 3months) will be obtained for each arm. And these differences will be compared between the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Said Saghieh, MD, Study Director — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No